CLINICAL TRIAL: NCT07084415
Title: Effect of Laser Acupuncture on Neck and Shoulder Pain in Lactating Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yara Mokhtar Abd El-Latif, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005732
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postural correction exercise group (Active Comparator): The participants will receive postural correction exercises for 10 repetitions, 5 sessions per week for 4 weeks.
  Interventions: Other: Postural correction exercise
- Postural correction exercise and laser acupuncture group (Experimental): The participants will receive postural correction exercises (10 repetitions, 5 sessions per week for 4 weeks.), and laser acupuncture for 7 minutes twice per week for 4 weeks.
  Interventions: Other: Postural correction exercise; Device: Laser acupuncture

INTERVENTIONS:
Other: Postural correction exercise — Each participant will be given cervical thoracic spine correction exercises in the form of thoracic Roll Stretching Exercises, shoulder Bracing (Shoulder Retraction), superman Pose, chin Tuck (Cervical Retraction), five days a week for 4 weeks
Device: Laser acupuncture — A dermatograph pencil (COLOURED®) will be used to draw circles with diameters of 2 cm around the application points. Each point will be stimulated for 30 seconds.
  The laser will be placed at the specific acupuncture points in shoulder and cervical regions.
  Each woman in the study group will be treated by laser acupuncture for 7 minutes twice a week for 4 weeks.
  Acupuncture points of the neck:
  B10 (Tianzhu), GB 20 (Fengchi), GB 21 (jianjing), and EX-HN15 (jianzhongsgu). Acupuncture points of shoulder: LI 14 (Binao), LI 15 (Jianyu), TE 14 (Jianlio), LI 4 (Hegu),LI16 (Jugu), ST 38 (Tiaoko), SI 10 (Naoshu),LI 11 (Quchi),TE 15 (Tianliao),LU 1 (Zhongfu),
  Parameter of laser:
  wavelength: 808[nm], Operating mode: Continuous wave, Output power: 100 [mW], Power density: 333[mW/cm], area irradiated:0.3 cm2, Total time per point: 30[s], Angle of application:90 degree.
  Arms: Postural correction exercise and laser acupuncture group

SUMMARY:
The purpose of this study is to investigate the effect of laser acupuncture on neck and shoulder pain in lactating women.

DETAILED DESCRIPTION:
Breastfeeding was the most common daily living activity that caused neck and shoulder pain to become worse in lactating women, the mother's position is a head-down position to maintain eye contact with the infant, so there are possibilities of breastfeeding-related neck pain .

It was revealed that neck and shoulder pain greatly influenced the health of postpartum women; it led to a reduction in the level of quality of life of postpartum women.

Acupuncture is a choice for therapeutic intervention of patients with neck and shoulder pain and can be incorporated into rehabilitation.

laser acupuncture (LA) uses a low-intensity, non-thermal laser irradiation to stimulate the acupoints. LA may improve pain, disability, and functional levels in musculoskeletal disorders like shoulder and neck pain

ELIGIBILITY:
Inclusion Criteria:

* Lactating women Suffering from cervical and shoulder pain.
* Their body mass index will be less than 30 kg/m².
* Primipara and multipara "2:3 times" women.
* six weeks to one year after childbirth.

Exclusion Criteria:

* Neurological disorders.
* Musculoskeletal disorders as cervical discopathy or shoulder impingement syndrome.
* History of cervical or shoulder surgery.
* Infection or malignancy.
* Take any medical treatment or physiotherapy interventions in the past one month.
* Fibromyalgia or myopathy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  The Visual analogue scale will be used to measure the pain intensity before and after the treatment program. The VAS is a 10-point scale comprising a number from 0 through 10; 0 indicates "no pain", and 10 indicates the "worst imaginable pain
Pressure pain threshold | 4 weeks
  The pressure algometer will be used to assess pressure pain threshold before and after treatment. The examiner will determine the main 6 points of assessment on each side of cervical and shoulder girdle areas:
  * 2 cm lateral to the cervical vertebrae 2 (C2) spinous processes.
  * At the middle point of the upper trapezius muscle (between C7 and the acromion).
  * At levator scapulae (2 cm superior to the superior angle of the scapulae).
  * At mid-line of deltoid muscle. Three consecutive measurements will be made, with an interval of 30 s between them, and the average value will be recorded.
cervical flexion range of motion | 4 weeks
  The patient will be in sitting position the head will be in 0-degree rotation or lateral flexion, stabilize shoulder girdle and chest by strap, The central fulcrum of goniometer will be in the external auditory meatus, the proximal arm is perpendicular, the distal arm with the base of the nares, The patient will be asked to flex her cervical until end of range. Normal cervical flexion range of motion is 80 degrees
cervical extension range of motion | 4 weeks
  The patient will be in sitting position the head will be in 0-degree rotation or lateral flexion, stabilize shoulder girdle and chest by strap, The central fulcrum of goniometer will be in the external auditory meatus, the proximal arm is perpendicular, the distal arm with the base of the nares, The patient will be asked toextend her cervical until end of range. Normal cervical extension range of motion is 50-70 degrees
cervical side bending | 4 weeks
  The patient will be in sitting position the head will be in 0 degree rotation or flexion or extension, stabilize shoulder girdle and chest by strap. The central fulcrum of goniometer will be over the spinous process of C7 vertebra, the proximal arm is align with spinous process of the thoracic verebrae ,the distal arm will align with dorsal of the head, the patient will be asked to side bend her cervical to end range. Normal range of motion of cervical side bending is 20-45 degrees.
cervical rotation | 4 weeks
  The patient will be in sitting position the head will be in neutral position, stabilize shoulder girdle and chest by strap, Center fulcrum of the goniometer over the center of the cranial aspect of the head, Align proximal arm parallel to an imaginary line between the two acromial processes, Align distal arm with the tip of the nose. If a tongue depressor is used, align the arm of the goniometer parallel to the longitudinal axis of the tongue depressor, The patient will be asked to rotate her cervical until end of range. Normal range of motion of cervical rotation is 70-90 degrees.
Shoulder flexion range of motion | 4 weeks
  The patient will be in supine lying position the knee will be 90-degree position, stabilize scapula and thorax girdle, Center fulcrum of the goniometer over the lateral aspect of the greater tubercle, Align proximal arm parallel to the midaxillary line of the thorax, Align distal arm with the lateral midline of the humerus. The patient will be asked to flex her shoulder until end of range.
  Normal range of motion of shoulder flexion is 150-180 degrees.
Shoulder extension range of motion | 4 weeks
  The patient will be in prone position, Center fulcrum of the goniometer over the lateral aspect of the greater tubercle, Align proximal arm parallel to the midaxillary line of the thorax, Align distal arm with the lateral midline of the humerus. The patient will be asked to extend her shoulder until end of range. Normal range of motion of shoulder flexion is 45-60 degrees.
Shoulder abduction range of motion | 4 weeks
  The patient will be in supine lying position., Center fulcrum of the goniometer close to the anterior aspect of the acromial process, Align proximal arm so that it is parallel to the midline of the anterior aspect of the sternum, Align distal arm with the anterior midline of the humerus, The patient will be asked to abduct her shoulder until end of range. Normal range of motion of shoulder flexion is 150 degrees.
Shoulder internal rotation range of motion | 4 weeks
  The patient will be in supine lying position, Center fulcrum of the goniometer over the olecranon process, Align proximal arm so that it is either perpendicular to or parallel with the floor, Align distal arm with the ulna, using the olecranon process and ulnar styloid for reference. The patient will be asked to internal rotate her shoulder until end of range. Normal range of motion of shoulder internal rotation is 70-90 degrees.
Shoulder external rotation range of motion | 4 weeks
  The patient will be in supine lying position, Center fulcrum of the goniometer over the olecranon process, Align proximal arm so that it is either perpendicular to or parallel with the floor, Align distal arm with the ulna, using the olecranon process and ulnar styloid for reference. The patient will be asked to internal rotate her shoulder until end of range. Normal range of motion of shoulder internal rotation is 90 degrees.

SECONDARY OUTCOMES:
Functional disability | 4 weeks
  Neck disability index will be used to assess functional disability before and after treatment. It consists of 10 questions: pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. 5 Each item is scored from 0 (no disability) to 5 (total disability). The maximum possible score is 50.
Shoulder and pain disability index (SAPDI) | 4 weeks
  It will be used to assess the degree of shoulder pain and discomfort in performing activities of daily living. It consists of 13 items divided into two subscales: 5 items for pain and 8 items for disability. The SPADI total score is the mean of the pain and disability sub-scores. Higher score indicates more disability.
Breastfeeding Self Efficacy assessment | 4 weeks
  It will be used to measure mother's confidence in her ability to breastfeed. The scale is a 14-item, self-administered instrument, where items are preceded by the phrase "I can always" and scored on a 5-point Likert scale ranging from 1 (not at all confident) to 5 (always confident). As such, total scores can range from 14 to 70, with higher scores reflecting greater levels of breastfeeding self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Hussein, Professor, Study Director — Al-Azhar University; Doaa Osman, Professor, Study Chair — Cairo University
Locations (1):
- Yara Mokhtar Abd El-Latif, Cairo, Egypt